CLINICAL TRIAL: NCT01530581
Title: A Randomized Multicentre Study Comparing G-CSF Mobilized Peripheral Blood and G-CSF Stimulated Bone Marrow in Patients Undergoing Matched Sibling Transplantation for Hematologic Malignancies
Brief Title: Study Comparing G-CSF Mobilized Peripheral Blood and G-CSF Stimulated Bone Marrow in Patients Undergoing Matched Sibling Transplantation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2081-076
Record Dates: First submitted 2012-01-23; First posted 2012-02-10 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Transplantation for Hematologic Malignancies

ARMS (2):
- G-BM Transplant (Experimental)
  Interventions: Procedure: G-BM Transplant
- G-PB Transplant (Other): G-PB Transplant
  Interventions: Procedure: G-PB Transplant

INTERVENTIONS:
Procedure: G-PB Transplant — G-PB Transplant
  Arms: G-PB Transplant
Procedure: G-BM Transplant — G-BM Transplant
  Arms: G-BM Transplant

SUMMARY:
This is a Randomized Multicentre study Comparing GCSF Mobilized Peripheral Blood and GCSF stimulated Bone Marrow in Patients undergoing matched sibling Transplantation for Haematologic Malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Recipient must

  1. Be between the ages of 16 and 65 years old
  2. Have one of the following hematologic malignancies:

     * Acute myeloid leukemia (de novo, secondary or therapy related) in untreated 1st relapse or in remission or with evidence of molecular relapse but blasts less than 5%
     * Chronic myeloid leukemia in chronic or accelerated phase (de novo or therapy related)
     * Myelodysplasia (de novo or therapy related)
     * Other hematologic malignancy (de novo or therapy related) including but not limited to: ALL (CR 1, CR2 or CR3), CLL, non-Hodgkin's lymphoma, Hodgkin's lymphoma
  3. Must be receiving a myeloablative conditioning regimen of busulfan and cyclophosphamide or TBI and cyclophosphamide or other myeloablative regimen approved by the Clinical Study Chair. (Regimens containing ATG are not allowed.)
  4. Have an HLA-identical sibling donor
  5. Meet the transplant centre's criteria for myeloablative allogeneic transplantation*
  6. Have an ECOG performance status of 0, 1 or 2
  7. Have given signed informed consent

Donor must

1. Be 18 years of age or older. (Upper age limit is at the discretion of the transplant physician at the collection centre.)
2. Be able to undergo general anesthesia and BM harvest or peripheral blood collection as per assessment by a transplant physician. (If an anesthetist assesses a donor after randomization and determines the donor should not undergo general anesthesia, then the donor and recipient will be withdrawn from the study.)
3. Be a sibling of the recipient
4. Be a 6/6 HLA match of the recipient. HLA typing is by serologic or DNA methodology for A and B and by DNA methodology for A and B and by DNA methodology for DRB1 (intermediate resolution)
5. Have given signed informed consent

Exclusion Criteria

Recipient

1. The recipient is HIV antibody positive

Donor

1. The donor is unable to undergo general anesthesia, bone marrow harvest or peripheral blood collection
2. The donor is pregnant or breastfeeding at the time of progenitor cell collection
3. The donor has a history of malignant disease within the last 5 years or current malignancy other than non-melanomatous in situ skin carcinoma or cervical carcinoma in situ
4. The donor is HIV antibody positive
5. The donor has a known sensitivity to E. coli-derived products
6. The donor and recipient are identical twins

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2008-11; Primary Completion 2012-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Efficacy | 2 years
  The use of G-BM is associated with a longer time to treatment failure (extensive chronic GVHD, relapse, death) than is the use of G-PB for adult myeloablative allogeneic transplantation for hematologic malignancies.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Al Jurf, MD, Principal Investigator — King Faisal Specialist Hospital & Research Center
Locations (1):
- King Faisal Specialist Hospital & Research Center, Riyadh, Saudi Arabia